CLINICAL TRIAL: NCT03931980
Title: Robotic Versus Laparoscopic Approach for Rectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Binh Dan Hospital (Other)
Responsible Party: Principal Investigator, NGUYEN PHUC MINH, Medical Doctor, Binh Dan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD012019
Record Dates: First submitted 2019-04-03; First posted 2019-04-30 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; robotic surgery; laparoscopic surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic surgery (Experimental): Patients undergoing robotic surgery for removal of rectal cancer.
  Interventions: Procedure: Robotic-assisted rectal cancer resection and Laparoscopic rectal cancer resection
- Laparoscopic surgery (Experimental): Patients undergoing laparoscopic for removal of rectal cancer
  Interventions: Procedure: Robotic-assisted rectal cancer resection and Laparoscopic rectal cancer resection

INTERVENTIONS:
Procedure: Robotic-assisted rectal cancer resection and Laparoscopic rectal cancer resection — we perform robotic surgery using the da Vinci Robot System Si version and laparoscopic surgery to treat rectal cancer
  Other Names: Laparoscopic rectal cancer resection; Da Vinci robotic system; Rectal cancer surgery; Robotic rectal cancer surgery

SUMMARY:
Colorectal cancer is a common malignancy in Viet Nam. Laparoscopic surgery becomes a standard treatment in many centers. Today, robotic surgery is a new option for treating colorectal cancer with some advantages such as magnified 3D view, precise movements.

Answer on safety and feasibility of robotic surgery for colorectal cancer are not available in Viet Nam. Therefore, the investigators conducted a study " Robotic versus Laparoscopic Approach for Rectal Cancer Surgery".

DETAILED DESCRIPTION:
Rectal cancer is a common surgical disease

ELIGIBILITY:
Inclusion Criteria:

* able to provide written informed consent
* Diagnosis of rectal cancer amenable to curative surgery by anterior resection, low anterior resection, ultra-low anterior resection, abdominal perineal resection, staged T1-T4a, N0-2, M0

Exclusion Criteria:

* Advanced cancer not amenable to curative surgery
* patient did not agree to participate in research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Conversion to open surgery | 1 day
  the rate of conversion to open surgery

SECONDARY OUTCOMES:
Time of surgery | 1 day
  Time of surgery on the robot compare to laparoscopic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hung V Tran, PhD, Study Director — Binh Dan Hospital
Locations (1):
- Binh Dan hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No